CLINICAL TRIAL: NCT04109495
Title: Usefulness of Smartphone Application for Improving Nutritional Status of Pancreatic Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1-2016-0061
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study designed to investigate the usefulness of the Noom smartphone application on nutrition management of pancreatic cancer patients. We randomly assigned patients with first diagnosed pancreatic cancer to Noom user group or non-Noom user group. A total of 40 participants were included for randomization. All patients underwent nutritional assessments (PG-SGA), laboratory test and quality of life assessments (EORTC QLQ) at enrollment, 4, 8, and 12 weeks. During study period, Noom user group voluntarily record meals and get feedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart phone application(NOOM) (Other)
  Interventions: Other: Smart phone application(NOOM)
- Non-user (Other)
  Interventions: Other: Non-user

INTERVENTIONS:
Other: Smart phone application(NOOM) — The study population included first diagnosis of pancreatic cancer patients within 3 months of pancreatic cancer center visit, and randomly assigned to the use of Noom user group and non-use group. A total of 40 patients, 20 from each group, were used to examine nutritional status(PG-SGA), blood index analysis, and quality of life(EORTC QLQ) at 0, 4, 8, and 12 weeks. At the same time, the patients voluntarily record meals and receive feedback using Noom. The purpose and contents of this study are explained in detail to the subjects, and written consent is obtained. The questionnaire items included gender, age, weight, type of diagnosed digestive disease, treatment method, nutritional supplement, oral status and intake of oral supplement foods, and past medical history. To assess the nutritional status using laboratory data, blood(about 8ml) is collected for each visit.
  Arms: Smart phone application(NOOM)
Other: Non-user — The patients dose not use Noom application. A total of 40 patients, 20 from each group, were used to examine nutritional status (PG-SGA), blood index analysis, and quality of life (EORTC QLQ) at 0, 4, 8, and 12 weeks. The purpose and contents of this study are explained in detail to the subjects, and written consent is obtained. The questionnaire items included gender, age, weight, type of diagnosed digestive disease, treatment method, nutritional supplement, oral status and intake of oral supplement foods, and past medical history. To assess the nutritional status using laboratory data, blood (about 8ml) is collected for each visit. At each visit, you will be assessed nutritional status and quality of life through the PG-SGA and EORTC QLQ.
  Arms: Non-user

SUMMARY:
Malnutrition of hospitalized patients is reported in the range of 20-60% according to the definition and assessment method of malnutrition.

In particular, the incidence of malnutrition in cancer patients is high up to 30-85%.

Gastrointestinal disease is related to the digestion and absorption of nutrition therefore malnutrition rate of those patients is relatively high. Careful management of nutrition support is needed.

Malnutrition causes dysfunction of the mesenteric membrane, immune function impairment, decreased function of major organs such as liver, kidney and heart and alteration in pharmacodynamics. It could also increase infection rate and complications of chemotherapy, delay recovery time, so that increase morbidity, mortality and length of hospital stay.

Proper nutrition management reduces malnutrition prevalence and medical costs of hospitalized patient, therefore nutrition screening and evaluation is necessary. The recent spread of smartphones has made it easier to record and evaluate meals, which are used in the diet market for weight loss through meal records and feedback based on smartphone applications. This approach is also expected to benefit patients with gastrointestinal cancer, where proper nutrition and feedback are important. In particular, pancreatic cancer, the worst intractable cancer of mankind, is digestive cancer with the most severe muscle mass reduction and nutritional deterioration after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1) Among patients with pancreatic cancer who visited Severance Hospital of Yonsei University

1. Patients who received the explanation from the investigator and agreed to the written consent of the subject
2. Men or Women aged 20 to 70

2) First diagnosed with pancreatic cancer within 3 months 3) Patients scheduled to undergo first-line chemotherapy after the diagnosis of pancreatic cancer

Exclusion Criteria:

1. Those who have or had a history of abdominal surgery within the past 1 year
2. Those who have an acute illness (pneumonia, sepsis, shock, etc.) and have an infection at the time of registration
3. chronic liver disease and chronic obstructive pulmonary disease
4. Patients with nutrient absorption disorder due to gastrointestinal mucosal diseases (ulcerative colitis, Crohn's disease, acute and chronic diarrhea, etc.)
5. Severe disease patients (heart failure, liver failure, kidney failure and hemodialysis, etc.)
6. Those who are pregnant or breastfeeding
7. Those who have used steroids within the last one month
8. Patients diagnosed of peritoneal seeding or suspected GI obstructive sign
9. Those who are already taking nutritional supplements

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

PRIMARY OUTCOMES:
PG-SGA(Patient-Generated Subjective Global Assessment) | 12 weeks
  A patient-generated subjective global assessment (PG-SGA) for oncology patients has been developed by Ottery. This tool has two sections-a medical history section that is completed by the patient, and a physical assessment section that is completed by nursing, medical, or dietetic staff. The medical history section includes additional questions regarding the presence of oncology nutrition impact symptoms.
EORTC Questionnaires - Quality of Life | 12 weeks
  The European Organization for Research and Treatment(EORTC) questionnaire was designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of 5 multiitem scales (physical, role, social, emotional and cognitive functioning) and 9 single items(pain, fatigue, financial impact, appetite loss, nausea/vomiting, diarrhea, constipation, sleep disturbance and quality of life).

SECONDARY OUTCOMES:
Skeletal muscle index change | 8 weeks
  Cross-sectional skeletal muscle area (SMA, cm2) at this level is highly correlated with total body skeletal muscle mass. Adjustment of SMA for height2 results in skeletal muscle index (SMI, cm2/m2), a measure for relative muscle mass. Using skeletal muscle index change we evaluated sarcopenia in pancreatic cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keum J, Chung MJ, Kim Y, Ko H, Sung MJ, Jo JH, Park JY, Bang S, Park SW, Song SY, Lee HS. Usefulness of Smartphone Apps for Improving Nutritional Status of Pancreatic Cancer Patients: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Aug 31;9(8):e21088. doi: 10.2196/21088. PMID 34463630